CLINICAL TRIAL: NCT05256563
Title: A Biomarker for Personalized Care in Post-stroke Spatial Neglect
Status: Active, not recruiting | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: N3760-P
Record Dates: First submitted 2022-02-15; First posted 2022-02-25 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Spatial Neglect; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Right brain stroke survivors: People with right brain stroke who are recruited to the study.

SUMMARY:
More than 30,000 Veterans are hospitalized for stroke each year, and in the critical first months of recovery, at least half are disabled by abnormal 3-D spatial function (spatial neglect). Their self-care, mobility, and ability to return home are severely limited.

DETAILED DESCRIPTION:
Spatial Neglect (SN)is an underdiagnosed stroke-related condition--and a specific core set of symptoms--Aiming Spatial Neglect-- may have a major adverse effect on outcome. These same symptoms may predict excellent response to spatial neglect therapy. The investigators seek to develop a biological parameter for treatment assignment. In this two-year study, the investigators will enroll 45 people with right brain stroke who are at high risk of SN. The investigators will examine clinical brain images, behavioral assessment and research brain images at baseline and recovery at 3 and 6 months after study entry.

ELIGIBILITY:
Inclusion Criteria:

* Stroke survivors >18 years
* 1-8 months post-stroke
* Can undergo testing and give informed consent

Exclusion Criteria:

* Other serious
* Chronic neurological disorders
* Evidence of other serious strokes
* Inability to undergo testing or give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: See Inclusion and Exclusion Criteria
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in functional ability for daily life tasks assessed on the FONE-FIM at 3 months | baseline to 3 months
  Functional performance of daily life tasks will be assessed with the FONE-FIM questionnaire. This variable assesses improvement between baseline and 3 months. The FONE-FIM has has a minimum score of 18 and a maximum score of 126, being 126 the maximum level of independence in daily life activities. Therefore, change can be 0-108 points.
SN severity at baseline | baseline
  Catherine Bergego Scale--an examiner-assessed measure of functional performance specific to SN. The score goes from 0 to 30 determining mild (0-10), moderate (11-20) or severe (21-30) spatial neglect.
Change in functional ability assessed by the Barthel Index at 3 months | baseline to 3 months
  Functional performance of daily life tasks will be assessed with the Barthel Index questionnaire. This is has a minimum score of 0 and a maximum score of 100, with100 the maximum amount of help a person might need to perform daily life activities. Therefore, change at 3 months can be 0-100 points.
Change in functional ability for daily life tasks assessed on the FONE-FIM at 6 months | baseline to 6 months
  Functional performance of daily life tasks will be assessed with the FONE-FIM questionnaire. This variable assesses improvement between baseline and 6 months. The FONE-FIM has has a minimum score of 18 and a maximum score of 126, being 126 the maximum level of independence in daily life activities. Therefore, change can be 0-108 points.
SN severity at 3 months | 3 months post-baseline
  Catherine Bergego Scale--an examiner-assessed measure of functional performance specific to SN. The score goes from 0 to 30 determining mild (0-10), moderate (11-20) or severe (21-30) spatial neglect.
SN severity at 6 months | 6 months post-baseline
  Catherine Bergego Scale--an examiner-assessed measure of functional performance specific to SN. The score goes from 0 to 30 determining mild (0-10), moderate (11-20) or severe (21-30) spatial neglect.
Change in functional ability assessed by the Barthel Index at 6 months | baseline to 6 months
  Functional performance of daily life tasks will be assessed with the Barthel Index questionnaire. This is has a minimum score of 0 and a maximum score of 100, with100 the maximum amount of help a person might need to perform daily life activities. Therefore, change at 6 months can be 0-100 points.

OTHER OUTCOMES:
Number of stroke survivors that have evidence of Aiming SN | baseline
  The investigators will examine whether or not stroke survivors have evidence of Aiming SN on validated measures such as the Computerized Line Bisection where the person must bisect lines using the computer mouse. This tests determines if the person has an aiming or where bias.

CONTACTS AND LOCATIONS:
Overall Officials: Anna M. Barrett, MD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/63/NCT05256563/ICF_000.pdf